CLINICAL TRIAL: NCT00002309
Title: A Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study of Azithromycin as Prophylaxis Against the Development of Mycobacterium Avium Complex Disease in HIV-Infected People
Brief Title: A Study of Azithromycin in the Prevention of Mycobacterium Avium Complex Disease (MAC) in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 058I; 066-155
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Azithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To evaluate the efficacy and safety of azithromycin administered once a week in the prevention of disseminated Mycobacterium avium complex (MAC) in severely immunocompromised HIV-infected patients with a CD4 count < 100 cells/mm3.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Anti-pneumocystis prophylactic therapy (dihydropteroate synthetase inhibitors with or without dihydrofolate reductase inhibitors, pentamidine).

Allowed:

* Concomitant anti-HIV therapy (AZT, ddI, ddC) or antifungal therapy (including azoles).

Patients must have:

* HIV infection.
* CD4 count < 100 cells/mm3.
* No MAC positive blood cultures within 1 month prior to study entry.
* No symptoms suggestive of disseminated MAC infection (including unexplained diarrhea, fever, and night sweats) within 1 month of study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Positive PPD within 3 months prior to study entry (negative PPD defined as < 5 mm induration).
* Chest x-ray suggestive of any active disease, in particular tuberculosis.
* Known hypersensitivity to macrolide antibiotics.
* Any other acute clinical condition likely to interfere with completion of the protocol.
* Inability to care for self without considerable assistance and medical care.

Concurrent Medication:

Excluded:

* Other investigational new drugs (except for foscarnet or ddC) unless prior agreement has been reached between the investigator and the Pfizer project physician.
* Concomitant putative immunostimulants.

Patients with the following prior conditions are excluded:

History of MAC or Mycobacterium tuberculosis (MTb) infection.

Prior Medication:

Excluded within the past 4 weeks:

* Any putative anti-MAC therapies including rifampin, rifabutin, clofazimine, ethambutol, cycloserine, ethionamide, amikacin, and ciprofloxacin or other quinolones thought to be active against MAC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - San Diego Naval Hosp, San Diego, California
  - Womack Army Med Ctr / Med Clinic, Fort Bragg, North Carolina
  - United States Air Force Med Ctr, Lackland Air Force Base, Texas

REFERENCES:
- [Background] Oldfield EC, Dickinson G, Chung R, Wallace MR, Craig DB, Fessel WJ, Joyce MP, Mckee KT, Melcher G, Wagner KF, Williams WJ, Zajdowicz M, Heifits L, Dunne MW, Berman J. Once weekly azithromycin for the prevention of Mycobacterium avium complex (MAC) infection in AIDS patients. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:90